CLINICAL TRIAL: NCT02265419
Title: Case-observation and Compassionate Use: Use of Extracorporeal Treatment With the Cytosorb-Adsorber for the Reduction of Postoperative Hyperinflammation and SIRS After Heart-surgery With the Use of a Heart-lung-machine
Brief Title: Use of Extracorporeal Treatment With the Cytosorb-Adsorber for the Reduction of SIRS in Heart Surgery Patients
Acronym: CASHSP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Rostock (Other)
Responsible Party: Principal Investigator, Dr. Martin Sauer, MD, PD Dr., University of Rostock
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A 2014-0064
Record Dates: First submitted 2014-10-09; First posted 2014-10-15 (Estimated); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Multiple Organ Failure
Keywords: hyperinflammation, Cytosorb
MeSH Terms: conditions — Multiple Organ Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cytosorb group (Experimental): Extracorporeal treatment with the Cytosorb adsorber for 24 hours after heart surgical operation.
  Interventions: Device: Extracorporeal treatment with the Cytosorb adsorber

INTERVENTIONS:
Device: Extracorporeal treatment with the Cytosorb adsorber — The extracorporeal treatment with the Cytosorb-Adsorber will be started 6 hours after heart surgery operation, the extracorporeal treatment duration will be 24 hours and the observation time 90 days.

SUMMARY:
Heart-surgery with the use of a heart-lung-machine can trigger the development of a full-blown SIRS (Systemic Inflammatory Response Syndrom) with multi organ failure and severe sepsis in the course of disease.

For the treatment of full-blown SIRS extracorporeal treatment like the Cytosorb-Adsorber are in clinical testing. The Cytosorb-Adsorber is a CE-signed medical device with approval for the treatment of severe sepsis and hyperinflammation. The adsorber remove not-specific cytokines and other inflammation mediators from the patients blood.

In this study (as a case-observation and compassionate use) the effect of extracorporeal treatment with the Cytosorb-Adsorber for the reduction of postoperative hyperinflammation and SIRS after heart-surgery with use of a heart-lung-machine will be observed.

The aim of the study is recording the influence of the treatment with the Cytosorb-Adsorber on the course of hyperinflammation and multi organ failure in comparison with a historic control group.

DETAILED DESCRIPTION:
All patients underlying heart surgery with the use of a heart-lung-machine and fullfilling of the inclusion-criteria should be sreened for the study. The study take place on two surgical intensive care units (PIT I and PIT II) of the university hospital Rostock, Germany. The extracorporeal treatment with the Cytosorb-Adsorber will be started 6 hours after end of the operation if written informed consent was obtained from all participants or from the patients' representatives if direct consent could not be received. The extracorporeal treatment duration will be 24 hours and the observation time 90 days.

The aim of the study is recording the influence of the treatment with the Cytosorb-Adsorber on the course of hyperinflammation and multi organ failure in comparison with a historic control group. The main-criterion is a significant difference in the mean-SOFA (Sequential Organ Failure Assessment)-score between the Cytosorb-group and the historic control group after 7 days. Beside criterions are the 30- and 90-day survival, time of respirator-therapy, length of ICU stay, severity of the Critical Illness Polyneuropathy and dosage of vasopressors on the days 1, 2 and 3.

From all patients basic demographic information, illness severity (APACHE II, SOFA scores), microbiological results, pre-morbidity, and clinical outcome for study cohort will recorded. At the days 1-4, 7, 14, 30 and before/after the extracorporeal treatment the patients will screened for clinical and immunological data: hemodynamic, inflammation, coagulation, hemolysis, temperature, organ function blood parameters and cytokines. "Day 1" was defined as the day of the beginning of the extracorporeal treatment. At days 1, 2 and 7 hemodynamic monitoring will done with the PiCCO-System (PULSION Medical Systems, Feldkirchen, Germany). For dynamic measurement of the liver function will used the LiMON-System (based on the indocyanin green plasma disappearance rate, PULSION) on the days 1, 2 and 7.

ELIGIBILITY:
Inclusion Criteria:

* After heart surgery with heart-lung-machine
* 2 or more positive SIRS criterions within 6 hours postoperative
* need of > 1,9 liter kristalloids within 6 hours postoperative
* centralvenous oxygen saturation >75% within 6 hours postoperative
* need of vasopressors (≥0,06 µg/Kg/Min) within 6 hours postoperative

Exclusion Criteria:

* Bleeding
* Thrombocyten < 20.000 /µl, INR>3,0
* HIV-Test positive
* Hepatitis C positive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2014-10; Primary Completion 2022-01 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
mean SOFA | day 7
  A significant difference in the mean-SOFA (Sequential Organ Failure Assessment)-score between the Cytosorb-group and the historic control group after 7 days.

SECONDARY OUTCOMES:
30- and 90-day survival | day 30, day 90
  Observation time 90 days.
time of respirator-therapy | day 90
  Observation time 90 days.
length of ICU stay | day 90
  Observation time 90 days.
dosage of vasopressors on the days 1, 2 and 3. | day 1, 2 and 3
  Use of Vasopressors are monitored.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Sauer, PD Dr., Principal Investigator — University of Rostock, University Hospital, Intensive Care, Schillingallee 35, 18055 Rostock, Germany
Locations (1):
- Intensive Care Units PIT 1+2, University hospital Rostock, Rostock, Germany